CLINICAL TRIAL: NCT05989581
Title: Treatment of American Heart Association/American College of Cardiology Stage 1 Hypertension in Pregnancy: A Randomized Control Trial
Brief Title: Chronic Hypertension and Pregnancy 2 (CHAP2) Pilot Project
Acronym: CHAP2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ayodeji Sanusi, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000010726
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Labetalol; Nifedipine

STUDY DESIGN:
Intervention Model Description: Patients with stage 1 HTN in pregnancy will be randomized to BP goals of <130/80mmHg or usual care to treatment only if BPs ≥140/90mmHg. For this pilot, the investigator will randomize a total of 74 eligible participants, 37 to active treatment to BP<130/80mmHg and 37 to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BP goal <130/80mmHg (Experimental)
  Interventions: Drug: Labetalol or Nifedipine
- BP goal <140/90 (usual care) (No Intervention)

INTERVENTIONS:
Drug: Labetalol or Nifedipine — The choice of anti-HTN will be based on the patient and provider's experience and preference. First line anti-HTN recommended in pregnancy- labetalol or nifedipine- will be administered to patients. At least weekly, a study team member will review the participants' BPs and, if randomized to intervention and a higher dose is needed to maintain BPs <130/80 mmHg, the study team member will communicate with the clinical team, led by a University of Alabama Maternal Fetal Medicine Attending, in order to ensure coordination between the research and clinical care teams. Labetalol will be initiated at 200 mg twice daily and escalated in 200mg /dose daily until BP<130/80mmHg to a maximum dose of 2400mg/day. Procardia will be initiated at 30mg XL once daily and uptitrated in 30mg increments until a maximum dose of 120mg daily. Postpartum, titration will occur in similar fashion. The patient will be transitioned to her primary care provider for BP management after the 6-week postpartum visit.
  Arms: BP goal <130/80mmHg

SUMMARY:
The CHAP2 study is designed to provide preliminary data for a larger multicenter study to assess whether treatment of stage 1 hypertension (HTN) in pregnancy improves maternal and or neonatal outcomes. The primary objective of this pilot study is to determine if anti-HTN treatment to BP<130/80mmHg in pregnant patients with stage 1 HTN is associated with a difference in birthweight percentile at delivery. Patients with stage 1 hypertension in pregnancy will be randomized to BP goals of <130/80mmHg or usual care to treatment only if BPs ≥140/90mmHg. For this pilot, the investigator will randomize a total of 74 eligible participants, 37 to active treatment to BP<130/80mmHg and 37 to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton gestation
* No fetal anomalies
* Blood pressures 130-139/80-89mmHg on two occasions at least 4 hours apart prior to 20 weeks gestation
* Planning to deliver at UAB Hospital
* No indication for pregnancy termination
* Receiving care at the UAB prenatal clinics

Exclusion Criteria:

* Declines Randomization
* Known diagnosis of chronic hypertension ( BP ≥ 140/90mmHg) or current antihypertensive medication use
* Fetal demise diagnosed prior to enrollment
* Known major structural of chromosomal abnormalities prior to enrollment
* Contraindication to first line antihypertensive (Nifedipine/ Labetalol)
* Comorbidities requiring BP goals < 130/80mmHg

Ages: 14 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal Birthweight percentile | at delivery of infant
  To determine whether anti-HTN treatment to BP<130/80mmHg in pregnant patients with Stage 1 HTN is associated with a difference in birthweight percentile at delivery

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No